CLINICAL TRIAL: NCT06942988
Title: Efficacy of Intracavernous Platelet-rich Plasma Injection in the Treatment of Erectile Dysfunction
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Collaborators: t-biyoteknoloji labaratuvar estetik medikal kozmetik san. ve tic. ltd. şti. (Unknown)
Responsible Party: Principal Investigator, Yavuz Onur Danacıoğlu, Medical Doctor, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICPRPforED
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Erectile Dysfunction
Keywords: platelet-rich plasma; Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ICPRPforED (Experimental): Patients were planned to receive 3 sessions of intracavernous PRP injection once a month. Patients will be evaluated with IIEF scores and their partners with FSFI scores before treatment, during each procedure and 3 months after treatment.
  Two tubes of venous blood (8 ml each) will be collected from the patient by phlebotomy into MEDEX PRP tube. PRP will be prepared with 2000rpm-2min protocol and all plasma will be collected. PRP (approximately 5cc) will be applied proximally and distally to the bilateral cavernous body of the penis. In order to decrease venous return and increase the effectiveness of platelets in the cavernous body, a tourniquet will be applied to the penis with a ring from the proximal side, wait 20 minutes and remove the tourniquet.
  Interventions: Biological: intracavernous platelet rich plasma therapy

INTERVENTIONS:
Biological: intracavernous platelet rich plasma therapy — intracavernous platelet-rich plasma therapy for erectile dysfunction

SUMMARY:
Investigation of the efficacy of autologous platelet-rich plasma administration on the potency of patients with vasculogenic and/or neurogenic erectile dysfunction

ELIGIBILITY:
Inclusion Criteria:

- 1)40-70 years old male, sexually active heterosexual, 2) Patients with a diagnosis of mild to moderate erectile dysfunction (IIEF score between 8-21) according to the International Index of Erectile Function (IIEF) for at least 3 months, 3) Patients who cannot achieve an erection despite peroral PDE5 inhibitor and intracavernous alprostadil injection therapy

Exclusion Criteria:

1. Patients with psychogenic erectile dysfunction, 2) Patients with a history of priapism, penile fracture, peyronie, penile curvature 3) Patients with a history of radical prostatectomy, 4) Patients with a history of major pelvic trauma, surgery, radiotherapy, 5) Patients with a history of malignancy affecting survival, 6) Patients with severe psychiatric illness that impairs adherence to treatment, 7) Patients with any bleeding disorder or on anti-aggregants/coagulants.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-12-29 (Actual); Primary Completion 2025-07-29 (Estimated); Study Completion 2025-07-29 (Estimated)

PRIMARY OUTCOMES:
IIEF | 6 months
  To observe the increase in the International Index of Erectile Function (IIEF) score after treatment compared to before treatment in patients.

SECONDARY OUTCOMES:
FSFI | 6 months
  To observe FSFI score increases in patients' partners before and after treatment using the Female Sexual Function Inventory (FSFI).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Bakırköy Sadi Konuk Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided